CLINICAL TRIAL: NCT04662879
Title: A Prospective Study of Algorithm-based Screening in Patients With Glycemically Defined New Onset Diabetes to Evaluate Risk for and Earlier Detection of Pancreatic Ductal Adenocarcinoma; Early Detection Initiative (EDI) for Pancreatic Cancer
Brief Title: Early Detection Initiative for Pancreatic Cancer
Acronym: EDI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pancreatic Cancer Action Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 466; STU25020081 (Other: Univo Institutional Review Board); ONC-15162 (Other: Contract Research Organization)
Record Dates: First submitted 2020-11-20; First posted 2020-12-10 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hyperglycemia; Diabetes Mellitus; Pancreas Ductal Adenocarcinoma
Keywords: New Onset Diabetes; Hyperglycemia; Diabetes Mellitus; Pancreatic Ductal Adenocarcinoma; ENDPAC score; Weight loss; Glycemically defined new onset diabetes
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Intervention Model Description: Post-enrollment consent
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Site) (Experimental): Two interventions are performed:
  1. Have Enriching New-onset Diabetes for Pancreatic Cancer (ENDPAC) score calculated, and if Score is >0,
  2. Have abdominal imaging performed.
  Interventions: Other: Enriching New-onset Diabetes for Pancreatic Cancer (ENDPAC) score; Other: Abdominal imaging
- Observation Arm (Site) (No Intervention): Passive follow-up by electronic medical record for study endpoints of pancreatic cancer diagnosis.

INTERVENTIONS:
Other: Enriching New-onset Diabetes for Pancreatic Cancer (ENDPAC) score — ENDPAC is a model to risk-stratify patients with new onset diabetes and hyperglycemia for PDAC. Score is calculated using i) age, ii) change, over past year, in body weight and iii) change, over past year, in glucose/HbA1c values obtained from the electronic medical record.
  Arms: Intervention Arm (Site)
Other: Abdominal imaging — Using computerized tomography (CT) scan or magnetic resonance imaging (MRI), if CT scan is contra-indicated, patients with a high ENDPAC score (>0) are approached for informed consent to participate in the imaging intervention. Imaging (CT scan) is performed at up to two time points, study baseline and approximately 3-9 months following the first imaging study.
  Arms: Intervention Arm (Site)

SUMMARY:
The Early Detection Initiative for Pancreatic Cancer is a multi-center prospective study to determine if algorithm-based screening in patients with glycemically defined new onset hyperglycemia and diabetes has the potential for earlier detection of pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
The Early Detection Initiative (EDI), is designed to prospectively evaluate the performance characteristics of the Enriching New-onset Diabetes for Pancreatic Cancer (ENDPAC) model to enrich glycemically defined new-onset diabetes for pancreatic cancer. The study will also determine with elevated ENDPAC score occurs at a clinically meaningful lead time (>/= 4 months) before pancreatic cancer diagnosis.

Eligible patients are identified and enrolled based on a first-time elevation in fasting blood glucose parameters or glycated hemoglobin (HbA1c) to the level indicating glycemically defined new-onset diabetes as derived from records in their EMR. At sites performing the Intervention component of the study, all enrolled participants will have the Enriching New-onset Diabetes for Pancreatic Cancer (ENDPAC) score calculated using age, body weight and glucose or glycated hemoglobin values in their EMR. Patients with high ENDPAC score (>0) are approached for informed consent to participate in up to two imaging studies by computerized tomography (CT) scan or magnetic resonance imaging (MRI). In addition to imaging, participants will be asked to complete a study questionnaire. At sites that do not perform the Intervention component of the study, participants will be identified, enrolled, and followed by EMR data only. All enrolled participants are followed for development of PDAC.

This study is performed at locations with broad (institutional) consent for use of patient EMR information for research studies. Passive follow-up by EMR will occur for three years following enrollment. Any patient that has declined participation in EMR-based research at the institution is not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have given institutional consent for minimal risk studies.
* Patient must be ≥50 and ≤85 years of age at the time of diagnosis [index date Parameters of Diabetes Mellitus (PDM)].
* Patient must have index weight and left-window weight values available in electronic medical record (EMR).
* Patient must have hyperglycemia and/or diabetes as one of the following (all glycemic parameters, except for HbA1c, must be measured in an outpatient setting):

A. Glycated hemoglobin (HbA1c) ≥ 6.5%

OR

B. Any (2) PDMs on consecutive (≤90 days between PDMs) or simultaneous testing:

* Fasting Blood Glucose (FBG) ≥126 mg/dl
* Glycated hemoglobin (HbA1c) ≥ 6.5%
* Random Blood Glucose (RBG) ≥200 mg/dl
* 2 hour Post Glucose (PG) ≥ 200mg (11.1 mmol/L) during oral glucose tolerance test (OGTT)

OR

C. Any one (1) PDM present followed by an anti- diabetes medication ≤90 days after the index PDM date

* Patient must have ≥1 glycemic parameter measured in the past 91-548 days prior to the index PDM date (Left Window) without meeting inclusion criteria A, B, or C.
* For Intervention Sites, patients must meet inclusion criteria A, B, or C ≤90 days prior to enrollment.

Exclusion Criteria:

* Patient has declined institutional consent for minimal risk studies.
* Patient must not have any known past history of hyperglycemia and/or diabetes as defined by inclusion criteria A, B, or C

  *Transient diabetes (e.g. gestational and steroid-induced) is not an exclusion.
* Patient must not be on ongoing active treatment for cancer, and/or carry a current diagnosis of any cancer (except non-melanoma skin cancer). Non-invasive cancer of any organ (carcinoma-in-situ/high grade dysplasia) is not an exclusion.

  *Ongoing work up for suspicion of pancreatic cancer is not an exclusion.
* Patient must not have had a definitive diagnosis of pancreatic cancer prior to index PDM date.
* Patient must not be on any anti-diabetes medications prior to index PDM date.
* Patient must not be on chronic or acute use of steroid medications ≤90 days prior to the index PDM date.

  *Allowed: Nasal, topical steroids, oral budesonide, ophthalmic
* Patient must not have had an intra-articular steroid injection ≤ 7 days prior to the index PDM date.
* Patient must have values available in the EMR to calculate the ENDPAC score.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8869 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Validate the ENDPAC model | Baseline and approximately every six months for up to three years
  Prospectively validate the ENDPAC model.
Quantify potentially clinically meaningful lead time for earlier detection of PDAC | Baseline and approximately every six months for up to three years
  Measure the duration from G-NOD to date of clinical diagnosis of PDAC.

SECONDARY OUTCOMES:
Evaluate the risk of PDAC in G-NOD | Baseline and approximately every six months for up to three years
  Estimate the risk of PDAC in G-NOD in the average risk population including potentially clinically meaningful lead time for earlier detection of PDAC.
Proportion of incidental findings on imaging | Baseline and imaging follow-up visit, up to 9 months
  Evaluate, on imaging at the time of G-NOD, the proportion with incidental findings including those that require clinical work-up.
Risk of PDAC by subgroups | Baseline and approximately every six months for up to three years
  Estimate the risk of PDAC in the study population by racial and ethnic groups.
Reasons consent for intervention was declined | Baseline and approximately every six months for up to five years
  Evaluate the reasons invited participants decline consent for imaging intervention.

OTHER OUTCOMES:
Stage of disease at PDAC diagnosis | Baseline and approximately every six months for up to three years
  Evaluate the distribution and stage of disease at the time of PDAC diagnosis in participants with and without study imaging.
Glycemic parameters for ENDPAC model | Baseline and approximately every six months for up to three years
  Compare original ENDPAC score model to the modified ENDPAC score in the proportion of PDAC captured and lead time.
ENDPAC model by subgroups | Baseline and approximately every six months for up to three years
  Evaluate the proportion of PDAC captured and distribution of lead time across racial and ethnic populations.
Depression and Anxiety as early indicators | Baseline visit
  Capture the proportion of PDAC with symptoms of depression and anxiety, and how early it occurs before clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Chari, MD, Study Chair — M.D. Anderson Cancer Center; Anirban Maitra, MBBS, Principal Investigator — M.D. Anderson Cancer Center; Bechien Wu, MD, Principal Investigator — Kaiser Permanente; Avinash Kambadakone-Ramesh, MD, FRCR, Principal Investigator — Massachusetts General Hospital; Ziding Feng, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Kaiser Permanente Southern California, Kaiser Permanente Research, Pasadena, California
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Sharma A, Kandlakunta H, Nagpal SJS, Feng Z, Hoos W, Petersen GM, Chari ST. Model to Determine Risk of Pancreatic Cancer in Patients With New-Onset Diabetes. Gastroenterology. 2018 Sep;155(3):730-739.e3. doi: 10.1053/j.gastro.2018.05.023. Epub 2018 Jun 11. PMID 29775599
- [Background] Sharma A, Smyrk TC, Levy MJ, Topazian MA, Chari ST. Fasting Blood Glucose Levels Provide Estimate of Duration and Progression of Pancreatic Cancer Before Diagnosis. Gastroenterology. 2018 Aug;155(2):490-500.e2. doi: 10.1053/j.gastro.2018.04.025. Epub 2018 Apr 30. PMID 29723506
- [Background] Chari ST, Leibson CL, Rabe KG, Ransom J, de Andrade M, Petersen GM. Probability of pancreatic cancer following diabetes: a population-based study. Gastroenterology. 2005 Aug;129(2):504-11. doi: 10.1016/j.gastro.2005.05.007. PMID 16083707
- [Background] Khan S, Safarudin RF, Kupec JT. Validation of the ENDPAC model: Identifying new-onset diabetics at risk of pancreatic cancer. Pancreatology. 2021 Apr;21(3):550-555. doi: 10.1016/j.pan.2021.02.001. Epub 2021 Feb 8. PMID 33583686
- [Background] Chen W, Butler RK, Lustigova E, Chari ST, Wu BU. Validation of the Enriching New-Onset Diabetes for Pancreatic Cancer Model in a Diverse and Integrated Healthcare Setting. Dig Dis Sci. 2021 Jan;66(1):78-87. doi: 10.1007/s10620-020-06139-z. Epub 2020 Feb 28. PMID 32112260
- [Derived] Chari ST, Maitra A, Matrisian LM, Shrader EE, Wu BU, Kambadakone A, Zhao YQ, Kenner B, Rinaudo JAS, Srivastava S, Huang Y, Feng Z; Early Detection Initiative Consortium. Early Detection Initiative: A randomized controlled trial of algorithm-based screening in patients with new onset hyperglycemia and diabetes for early detection of pancreatic ductal adenocarcinoma. Contemp Clin Trials. 2022 Feb;113:106659. doi: 10.1016/j.cct.2021.106659. Epub 2021 Dec 23. PMID 34954100
- See also: Pancreatic Cancer Action Network Early Detection Initiative — https://www.pancan.org/research/early-detection-initiative/